CLINICAL TRIAL: NCT00914511
Title: A Phase I, Single-Center, Open-Label, Non-Randomized, Two-Cohort Study to Assess the Effect of Age on the Pharmacokinetics of Avanafil And To Determine Avanafil Semen Exposure and the Acute Effect of Avanafil on Sperm Function in Healthy Young Male Subjects Following a Single Oral Dose of 200 mg
Brief Title: A Pharmacokinetic Study of Avanfil in Healthy Young Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VIVUS LLC (Industry)
Responsible Party: Wesley Day, VP Clinical Development, Vivus, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: TA-014
Record Dates: First submitted 2009-06-03; First posted 2009-06-05 (Estimated); Last update posted 2011-01-07 (Estimated); Status verified 2011-01

CONDITIONS: Avanfil ADME; Semen Exposure; Sperm Function
Keywords: Semen; Sperm; Avanafil; Pharmacokinetics; Elderly
MeSH Terms: interventions — avanafil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy young males (Experimental): Healthy young males age 18-45, inclusive
  Interventions: Drug: avanafil 200mg
- Elderly males (Experimental): Elderly males 65 years of age and older
  Interventions: Drug: avanafil 200mg

INTERVENTIONS:
Drug: avanafil 200mg — single dose tablet of 200mg avanafil
  Arms: Healthy young males
Drug: avanafil 200mg — single tablet dose of 200mg avanafil
  Arms: Elderly males

SUMMARY:
The purposes of this study are to:

* Determine the effect of the study drug on sperm and semen of healthy young male subjects.
* Determine the effect of age on the amount of study drug in the blood of healthy subjects
* Learn about the safety of the study drug.
* Learn how subjects tolerate the study drug.

DETAILED DESCRIPTION:
This single-center, open-label, non-randomized, two-cohort, single-dose pharmacokinetic study will be conducted at a single site in the United States, in which at least 18 young (18-45 years, inclusive) male subjects in Cohort A and 14 elderly (65 years or older) males in Cohort B will be enrolled and dosed to achieve a total of at least 14 completed young subjects and 12 elderly subjects. Seminal fluid and plasma will be collected from Cohort A, whereas only plasma samples will be collected from Cohort B.

ELIGIBILITY:
Inclusion Criteria:

* Cohort A: Adult male subjects of 18 to 45 years of age inclusive Cohort B: Adult male subjects at least 65 years of age
* All subjects must be medically healthy with no clinically significant screening results.
* Male subjects should be willing to use a condom and spermicide during sexual activity for 90 days after last dosing of Avanafil and be willing to not donate sperm for 90 days after dosing.

Exclusion Criteria:

Major exclusion criteria for all subjects include:

* History or clinical evidence of clinically relevant cardiovascular (including thromboembolic disorders), hepatic, renal, hematologic, endocrine, pulmonary, gastrointestinal, psychiatric or neurological impairment
* Any clinically significant laboratory abnormalities as judged by the investigator
* Systolic blood pressure < 90 or >150 mmHg
* Diastolic blood pressure < 50 or > 95 mmHg
* Allergy to or previous adverse events with PDE5 inhibitors
* Use of prescription or over-the-counter drugs that are known to interfere with metabolism by the cytochrome P450 3A4 enzyme within 30 days of screening
* Use of any investigational drug within 30 days of screening
* Use of any prescription or over-the-counter drugs or herbal remedies within 14 days of screening
* History of alcohol or drug abuse within 18 months, history of smoking within 6 months
* Positive urine alcohol test
* Positive urine drug screen
* Positive urine cotinine test, positive serology for HIV, HCV, HBsAg
* Young males who have undergone vasectomy cannot participate in this-study
* Additional exclusion criteria are listed in Section 4.2.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-05; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Plasma pharmacokinetic parameters of avanafil and its metabolites will be evaluated including AUC (0-t), AUC(0-inf), Cmax, fu, t1/2, and tmax; Sperm motility, function and morphology; Avanafil exposure in seminal fluid | pre-dose (baseline) through 24 hours post-dose

SECONDARY OUTCOMES:
adverse events (each study visit); laboratory evaluations; electrocardiogram and physical examination; vital signs will be assessed at various times during the study. | pre-dose (baseline) through 24 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Shiyin Yee, PhD, Study Director — VIVUS LLC
Locations (1):
- MDS Pharma Services, Tempe, Arizona, United States